CLINICAL TRIAL: NCT01811797
Title: A Prospective, Randomized, Double Blind With Sham Control, Clinical Study to Assess the Safety and Efficacy Associated With Treating Patients Suffering From Erectile Dysfunction With Low Intensity Shockwaves by Renova
Brief Title: Safety and Efficacy Associated With Treating Erectile Dysfunction Patients With Low Intensity Shockwaves by Renova
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Initia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RENO-03-ICH
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Vasculogenic Erectile Dysfunction
Keywords: Erectile Dysfunction; Extracorporeal shockwave; Low intensity shockwaves
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Intensity Shockwave treatment (Experimental): 4 weekly sessions of Low Intensity Shockwave treatment.
  Interventions: Device: Low Intensity Shockwave by Renova
- Control group (Sham Comparator)
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Low Intensity Shockwave by Renova
  Arms: Low Intensity Shockwave treatment
Device: Sham treatment — Sham treatment that looks, sounds and feels like the real LISW treatment.
  Arms: Control group

SUMMARY:
This is a prospective, randomized, double-blind clinical study comparing safety and efficacy of the treatments performed with the Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT) device - "Renova" on symptomatic ED patients to the safety and efficacy of the control sham patients.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Vascular ED for at least 6 months
* International Index of Erectile Function 6 (IIEF-EF) between 11 to 25
* Positive response to PDE5-I (able to penetrate on demand=Responders)
* Negative response to PDE5-I (unable to penetrate on demand even with maximum PDE5-I dosage = Non-responders)
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Hormonal, neurological or psychological pathology
* Past radical prostatectomy or extensive pelvic surgery
* Recovering from cancer during last 5 years
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Past radiotherapy treatment of the pelvic region
* International normalized ratio (INR) > 3 for patients using blood thinners (such as Coumadin)

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the IIEF-EF (International Index of Erectile Function- Erectile Function Domain) score at 3 and 6 months post treatment | 1, 3 and 6 months post treatment

SECONDARY OUTCOMES:
Change from baseline in the SEP (Sexual Encounter Profile) Questions 2 and 3 at 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Change from baseline in the GAQ (Global Assessment Questions) at 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Change from baseline in the EDITS (Erectile Dysfunction Inventory of Treatment Satisfaction) score at 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Change from baseline in the Partner EDITS (Erectile Dysfunction Inventory of Treatment Satisfaction) score at 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Change from baseline in the IPSS (International Prostate Symptom Score) at the end of the treatment | 0 and 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209